CLINICAL TRIAL: NCT00635414
Title: An Open, Randomized, Two-way Crossover Study Comparing the Effect of 40mg Esomeprazole Administered Orally and Intravenously as a 15 Minute Infusion on Basal and Pentagastrin-Stimulated Acid Output in Subjects With Symptoms of Gastroesophageal Reflux Disease (GERD).
Brief Title: Open, Randomized, Two Way Crossover 40mg, Orally and Intravenously
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SH-NEP-0011; D9615C00011
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: GERD
Keywords: Gastroesophageal Reflux Disease (GERD), esomeprazole, Nexium
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

ARMS (2):
- 1 (Experimental): 40mg administered orally
  Interventions: Drug: Esomeprazole
- 2 (Experimental): 15 minute intravenous infusion
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — 40mg oral
  Other Names: Nexium
  Arms: 1
Drug: Esomeprazole — 15 minute intravenous infusion
  Other Names: Nexium
  Arms: 2

SUMMARY:
This study looks at the effect on basal and pentagastrin-stimulated acid output of 40 mg Esomeprazole (Nexium) administered orally and intravenously as a 15-minute infusion to people with symptoms of Gastroesophageal Reflux Disease (GERD)

ELIGIBILITY:
Inclusion Criteria:

1. Heartburn on at least 2 days of the past 7 days prior to screening, with or without a history of EE or a documented diagnosis of GERD within 6 months prior to screening, with or without a history of EE.
2. Body mass index (BMI) of ≥18.5 and ≤35 kg/m2. [BMI will be calculated using the following formula: weight (kg)/height (m)2.]
3. Able to communicate with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. History of esophageal, gastric, or duodenal surgery, except for simple closure of an ulcer.
2. History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.
3. Any significant "alarm symptoms", within the past 6 months, such as, unintentional weight loss, gastrointestinal bleeding, jaundice or any other sign indicating serious or malignant disease.
4. Abnormal lab test results, as indicated in the protocol.
5. Other diseases, as indicated in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-08; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
The maximal acid output (MAO) during pentagastrin stimulation after 10 days administration of 40 mg esomeprazole for both study periods. | MAO will be assessed after 10 days of treatment (Day 11 or Day 20)

SECONDARY OUTCOMES:
Basal acid output (BAO) after 10 days administration of 40 mg esomeprazole for both study periods. (Day 11 or Day 20) | BAO will be assessed after 10 days of treatment
To compare MAO when switching (after Day 2 in the second study period versus after Day 10 in the first study period) from oral to intravenous dosing and from intravenous to oral dosing. | Assessments at Day 2 and after Day 10 (Day 11 or Day 20)
To evaluate the safety of intravenous esomeprazole in subjects with symptoms of GERD. | Safety assessments throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca